CLINICAL TRIAL: NCT03306589
Title: An Open Label Parallel Group Study to Investigate the Optimum Methodology for the Use of LPS or GM-CSF as Challenge Agents on Healthy Participants by Assessing Inflammatory Biomarkers in Cantharidin-induced Skin Blisters, Peripheral Blood, and Urine
Brief Title: Lipopolysaccharide (LPS) or Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) Challenge Study on Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 207654
Record Dates: First submitted 2017-07-11; First posted 2017-10-11 (Actual); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Arthritis, Rheumatoid
Keywords: Inflammation; GM-CSF; LPS; Skin blisters; Healthy subjects; cantharidin
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation; Blister | interventions — Cantharidin; Lipopolysaccharides; Granulocyte-Macrophage Colony-Stimulating Factor; Saline Solution

STUDY DESIGN:
Intervention Model Description: Subjects in 2 separate groups will be randomized to receive either LPS or GM-CSF at the same time.
Masking Description: This will be an open label study and no masking will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Subjects receiving LPS: Part I and Part II (Experimental): Eligible subjects will be randomized to receive LPS in a dose-escalation manner ranging from 0.5 nanogram (ng)/kg to 4 ng/kg. Subjects will be hydrated prior to administration of LPS with normal saline at a rate of 250 mL/hour for 4 hours prior to dosing and 8 hours after dosing.
  Interventions: Biological: Cantharidin; Biological: Lipopolysaccharide; Drug: Saline Solution
- Subjects receiving GM-CSF: Part I and Part II (Experimental): Eligible subjects will be randomized to receive GM-CSF in a dose-escalation manner ranging from 5 to 15 microgram (µg)/kg.
  Interventions: Biological: Cantharidin; Biological: Granulocyte-Macrophage Colony-Stimulating Factor

INTERVENTIONS:
Biological: Cantharidin — 5 microliter (µL) of 0.2 percent Cantharidin solution (diluted in acetone) will be applied to all subjects on forearm by topical route.
Biological: Lipopolysaccharide — 0.5 to 4 ng/kg body weight of LPS formulated as suspension in normal saline will be administered to randomized subjects via intravenous (IV) route in dose-escalation manner.
  Arms: Subjects receiving LPS: Part I and Part II
Biological: Granulocyte-Macrophage Colony-Stimulating Factor — 5 to 15 µg/kg of GM-CSF will be administered to randomized subjects via subcutaneous (SC) route in the abdominal region in dose-escalation manner.
  Arms: Subjects receiving GM-CSF: Part I and Part II
Drug: Saline Solution — 0.9 percent sodium chloride will be administered via IV route to all subjects at a rate of 250 mL/hour for 4 hours prior to dosing with LPS and 8 hours after dosing with LPS.
  Arms: Subjects receiving LPS: Part I and Part II

SUMMARY:
This exploratory study aims to assess exposure of healthy subjects to systemic challenge with either LPS or GM-CSF. This will be done by measuring inflammatory mediators and cellular activation markers both in circulation and in skin blisters induced by exposure to cantharidin (an agent that causes blisters). LPS is often used to induce inflammation whereas GM-CSF is a cytokine and a key mediator in inflammatory diseases. In this 2 parts study, subjects will have 2 sessions in each part. Part I of the study is a dose-exploration phase and part II will be a continuation phase to draw more precise outcomes. In session 1, subjects will be randomized to receive either LPS or GM-CSF and will have 2 blisters induced on each forearm followed by blood draws and a blister harvest on each forearm at 24 and 48 hours post-induction. After a minimum of 14 days blister healing period, subjects will return for session 2. In part I, Up to 6 cohorts will be tested and all cohorts will have 2 sessions. For Part I, initially Cohort 1 will proceed with session 1. After their blister healing period, Cohort 1 will return for their session 2 visit in two groups (Group A and Group B) on different days. Group A will be dosed on the same day (one with LPS and one with GM-CSF) and Group B will be dosed on a different day (one with LPS and one with GM-CSF) after group A. Dose-escalation in Cohort 2-6 will be continued until the well tolerated dose has been determined. The same dose will be administered to an additional Cohort in Part II and the same 2-session design will be used. Approximately 24-30 healthy subjects will be enrolled for the study and the total duration of the study for each subject will be approximately 13 weeks from screening to follow up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 45 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by medical evaluation including: medical history, physical examination, laboratory tests, and electrocardiogram (ECG).
* Body mass index (BMI) within the range 19.0-30.0 kilogram per meter square (kg/m^2) (inclusive).
* All male subjects. All subjects must agree to use contraception during session 2 and refrain from donating sperm from session 2 to end of study (follow up 2 visits).
* Capable of giving signed informed consent.

Exclusion criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for human immuno deficiency virus (HIV) antibody.
* Persistent abnormal C-reactive protein/ white cell count (CRP/ WCC) levels at screening.
* Abnormal liver function tests at screening. For healthy subjects: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and bilirubin more than or equal to 1.5xupper limit of normal (ULN) (isolated bilirubin more than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35 percent) at screening.
* A positive pre-study drug/alcohol screen.
* Current, or chronic history of (h/o): liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), anaphylaxis, and /or anaphylactoid (resembling anaphylaxis) reactions; Cardiac, respiratory or renal disease (childhood asthma can be included); Sensitivity or severe allergic responses to any of the challenge agents or cantharidin, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation; Vasovagal syncope; Surgery or significant trauma in 3 months leading to study enrolment; Relevant skin conditions (for example recent h/o eczema or recurrent eczema, keloid, skin allergies, psoriasis, atopic dermatitis, and vitiligo) which in the opinion of the investigator could pose safety issues or cause interference with study procedures; Sepsis or known coagulation disorders; Peripheral edema, lymphangitis, lymph edema, pleural or pericardial effusion; Respiratory conditions including but not limited to asthma, Chronic obstructive pulmonary disease (COPD), and bronchiectasis and any current respiratory infection.
* Presence on either forearm of tattoos, naevi, hypertrophic scars, keloids, hyper or hypo-pigmentation. Subjects with very fair skin, very dark skin, excessive hair or any skin abnormalities that may, in the opinion of the Investigator, interfere with study assessments.
* Unable to refrain from the use of prescription drugs taken on an intermittent (as needed) basis or non-prescription drugs; these include non-steroidal anti-inflammatory drugs (NSAIDs), vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to Day 1 of session 1 and continuing until the final follow up visit).
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) or currently in a study of an investigational device.
* Previous exposure to LPS in a clinical research setting. Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within a 56-day period; Current smoker or former regular smoker within 6 months before the screening visit; Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study aimed to assess 2 models of systemic inflammatory response: exposure of healthy participants to systemic challenge with either Lipopolysaccharide (LPS) or Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF).
Pre-assignment Details: Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Groups:
- Part 1: LPS 0.5 ng/kg: Participants were randomized to receive 0.5 nanogram/kilogram (ng/kg) LPS as intravenous injection. After administration of LPS participant had two blisters induced on each arm followed by blood sample collection.
- Part 1: LPS 0.75 ng/kg: Participants were randomized to receive 0.75 ng/kg LPS as intravenous injection. After administration of LPS participant had two blisters induced on each arm followed by blood sample collection.
- Part 1: LPS 1 ng/kg: Participants were randomized to receive 1 ng/kg LPS as intravenous injection. After administration of LPS participant had two blisters induced on each arm followed by blood sample collection.
- Part 1: GM-CSF 60 µg/m^2: Participants were randomized to receive 60 microgram per meter square (µg/m^2) GM-CSF IV infusion. After administration of GM-CSF participant had two blisters induced on each arm followed by blood sample collection
- Part 2: Participants With LPS: Participants were planned to be dosed with LPS (0.5 with possible escalation up to 4 ng/kg) during Part 2 of the study.
- Part 2: Participants With GM-CSF: Participants were planned to be dosed with GM-CSF (60 to a maximum of 480 µg/m^2) during Part 2 of the study.
Period: Part 1 (69 Days)
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2 | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Started | 2 | 4 | 2 | 4 | 0 | 0
Completed | 2 | 4 | 2 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (69 Days)
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2 | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Started | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2 | Part 2: Participants With LPS | Part 2: Participants With GM-CSF | Total
Number analyzed (Participants) | 2 | 4 | 2 | 4 | 0 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.5 (4.95) | 35.5 (7.55) | 31.5 (10.61) | 33.5 (7.33) |  |  | 32.2 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 |  |  | 0
  Male | 2 | 4 | 2 | 4 |  |  | 12
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  White: WHITE/CAUCASIAN/EUROPEAN HERITAGE | 2 | 4 | 2 | 4 |  |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Baseline Primary Soluble Inflammatory Mediators in Blood: Tumor Necrosis Factor (TNF) Alpha and Interleukin (IL) 6 for LPS Arm
Description: Blood samples were collected at indicated timepoints for the analysis of primary soluble inflammatory mediators like TNF-alpha and IL-6 in blood. Latest pre-challenge LPS assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Each session was for three days. NA indicates that data was not available as standard deviation could not be calculated for a single participant. All participants who were randomized to receive the treatment (LPS or GM-CSF challenge) and received one dose of challenge agent were included in Safety Population.
Time Frame: Baseline, Session 2: -5, 10, 25, 40 minutes, 1 hour 10 minutes, 1 hour 40 minutes, 2 hours 40 minutes,5 hours 40 minutes on Day 1. Pre-fluid sample on Day 2 and Day 3
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Groups:
- Part 1: LPS 0.5 ng/kg: Participants were randomized to receive 0.5 ng/kg LPS as intravenous injection. After administration of LPS participant had two blisters induced on each arm followed by blood sample collection.
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg
Number analyzed (Participants) | 2 | 4 | 2
Picograms per milliliter
  IL-6, Session2,Day1, -5 minutes, n=2, 4, 2 | 2.4086 (0.09467) | 0.2798 (0.12546) | -0.0126 (0.01785)
  IL-6, Session2,Day1, 10 minutes, n=2, 4, 2 | 3.6460 (2.68681) | 0.2450 (0.16048) | 0.0123 (0.01746)
  IL-6, Session2,Day1, 25 minutes, n=1, 4, 2: number analyzed (Participants) | 1 | 4 | 2
  IL-6, Session2,Day1, 25 minutes, n=1, 4, 2 | 3.3141 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | 1.3623 (0.88290) | 1.8854 (0.15615)
  IL-6, Session2,Day1, 40 minutes, n=2, 4, 2 | 10.8074 (9.22779) | 8.7622 (8.41234) | 11.8672 (3.39867)
  IL-6, Session2,Day1, 1 hour 10 minutes, n=2, 4, 2 | 30.6395 (26.77767) | 81.0629 (104.23961) | 51.8232 (22.59507)
  IL-6, Session2,Day1, 1 hour 40 minutes, n=2, 4, 2 | 41.3221 (35.42047) | 193.7107 (218.97996) | 65.5675 (36.08430)
  IL-6, Session2,Day1, 2 hour 40 minutes, n=2, 4, 2 | 23.9321 (21.46574) | 133.2063 (92.47028) | 32.3842 (25.56374)
  IL-6, Session2,Day1, 5 hour 40 minutes, n=2, 4, 2 | 5.6991 (0.68051) | 2.5645 (1.20737) | 4.5141 (2.09962)
  IL-6, Session2,Day2, Pre-fluid sampling, n=2, 4, 2 | 17.8308 (16.52950) | 3.2880 (2.52703) | 0.3442 (0.03336)
  IL-6, Session2,Day3, Pre-fluid sampling, n=2, 4, 2 | -0.4610 (0.08488) | 0.5909 (0.96127) | 0.1542 (0.21529)
  TNF alpha, Session2,Day1, -5 minutes, n=2, 4, 2 | -0.2541 (0.33782) | -0.0726 (0.14769) | 6.4056 (8.96887)
  TNF alpha, Session2,Day1, 10 minutes, n=2, 4, 2 | 6.5720 (1.84896) | 2.3784 (2.45156) | 12.7647 (13.08048)
  TNF alpha, Session2,Day1, 25 minutes, n=1, 4, 2: number analyzed (Participants) | 1 | 4 | 2
  TNF alpha, Session2,Day1, 25 minutes, n=1, 4, 2 | 20.2469 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | 56.6529 (51.91815) | 84.6080 (33.94449)
  TNF alpha, Session2,Day1, 40 minutes, n=2, 4, 2 | 52.1665 (37.61641) | 157.5403 (165.48643) | 152.9415 (60.31144)
  TNF alpha, Session2,Day1, 1hour 10minutes, n=2,4,2 | 43.4949 (30.81434) | 202.6136 (215.34410) | 115.6693 (54.14279)
  TNF alpha, Session2,Day1, 1hour 40minutes, n=2,4,2 | 34.3031 (20.26768) | 147.3472 (122.68010) | 78.4734 (38.13965)
  TNF alpha, Session2,Day1, 2hour 40minutes, n=2,4,2 | 22.5571 (11.11988) | 68.8879 (24.42514) | 44.3372 (22.32753)
  TNF alpha, Session2,Day1, 5hour 40minutes, n=2,4,2 | 5.0087 (2.65663) | 15.4828 (7.05404) | 11.1378 (4.74317)
  TNF alpha, Session2,Day2,Pre-fluid sample, n=2,4,2 | 12.9279 (16.96994) | 1.2532 (0.83802) | 0.6475 (0.28268)
  TNF alpha, Session2,Day3,Pre-fluid sample, n=2,4,2 | 0.2453 (0.29126) | 0.2951 (0.39912) | 0.1391 (0.15747)

2. Primary Outcome: Part 1: Change From Baseline in Primary Soluble Inflammatory Mediators : Urinary Tetranor Prostaglandin D Metabolite (PGDM) LPS Arm
Description: The post-challenge urine samples were collected during session 2 after LPS challenge. In session 2, participants were encouraged to pass urine immediately before LPS challenge dose and urine voids were collected from after LPS until 12 hours post-LPS and the time of the urine collection were recorded as post-challenge 1 to 11. These samples were collected for measurement of tetranor-PGDM. Latest pre-challenge LPS assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. The data for normalized Tetranor PGDM was normalized by (Tetranor PGDM [pg/mL] divided by Creatinine [milligram per deciliter]) multiplied by 100. NA indicates that data was not available as standard deviation could not be calculated for a single participant.
Time Frame: Baseline, Session 2 Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Picograms per milligram
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg
Number analyzed (Participants) | 2 | 4 | 2
Picograms per milligram
  Session2, Day1,Post challenge1, n=2, 4, 2 | 73.846 (116.0073) | -85.080 (226.4168) | 134.806 (166.6716)
  Session2, Day1,Post challenge 2, n=2, 4, 2 | 99.438 (112.5337) | 88.984 (155.1855) | 276.788 (134.7190)
  Session2, Day1,Post challenge 3, n=2, 4, 2 | 32.006 (88.2367) | 25.390 (181.8009) | 200.337 (183.9484)
  Session2, Day1,Post challenge 4, n=2, 4, 2 | -119.091 (304.0503) | -68.209 (262.6169) | 140.482 (108.7880)
  Session2, Day1,Post challenge 5, n=1, 4, 2: number analyzed (Participants) | 1 | 4 | 2
  Session2, Day1,Post challenge 5, n=1, 4, 2 | 112.355 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | -146.294 (165.8587) | 184.263 (262.9020)
  Session2, Day1,Post challenge 6, n=0, 4, 1: number analyzed (Participants) | 0 | 4 | 1
  Session2, Day1,Post challenge 6, n=0, 4, 1 |  | -202.918 (197.6455) | -125.839 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Session2, Day1,Post challenge 7, n=0, 4, 1: number analyzed (Participants) | 0 | 4 | 1
  Session2, Day1,Post challenge 7, n=0, 4, 1 |  | -227.544 (226.2006) | 6.336 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Session2, Day1,Post challenge 8, n=0, 3, 1: number analyzed (Participants) | 0 | 3 | 1
  Session2, Day1,Post challenge 8, n=0, 3, 1 |  | -144.855 (53.7768) | -117.672 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Session2, Day1,Post challenge 9, n=0, 2, 1: number analyzed (Participants) | 0 | 2 | 1
  Session2, Day1,Post challenge 9, n=0, 2, 1 |  | -147.066 (39.8858) | -30.861 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Session2, Day1,Post challenge 10, n=0, 1, 1: number analyzed (Participants) | 0 | 1 | 1
  Session2, Day1,Post challenge 10, n=0, 1, 1 |  | -172.982 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | -37.732 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Session2, Day1,Post challenge 11, n=0, 1, 1: number analyzed (Participants) | 0 | 1 | 1
  Session2, Day1,Post challenge 11, n=0, 1, 1 |  | -199.316 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | -78.792 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

3. Primary Outcome: Part 2: Change From Baseline Primary Soluble Inflammatory Mediators in Blood: TNF Alpha and IL 6: LPS Arm
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of primary soluble inflammatory mediators like TNF-alpha and IL-6 in blood. Latest pre-challenge LPS assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Time Frame: Baseline, Session 2: -5, 10, 25, 40 minutes, 1 hour 10 minutes, 1 hour 40 minutes, 5 hours 40 minutes on Day 1. Pre-fluid sample on Day 2 and Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS
Number analyzed (Participants) | 0

4. Primary Outcome: Part 2: Change From Baseline Primary Soluble Inflammatory Mediators : Urinary Tetranor PGDM: LPS Arm
Description: Urine samples were planned to be collected for analysis. Latest pre-challenge LPS assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Time Frame: Baseline, Session 2 Day 1
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS
Number analyzed (Participants) | 0

5. Primary Outcome: Part 1: Change From Baseline in White Blood Cell Numbers in Blood: GM-CSF
Description: Blood samples were collected at indicated time-points for analysis of white blood cells. Latest pre-challenge GM-CSF assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Time Frame: Baseline, Session 2: 40 minutes, 2 hours 40 minutes, 5 hours 40 minutes, 9 hours 40 minutes on Day 1. Pre-fluid sample on Day 2 and Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Groups:
- Part 1: GM-CSF 60 µg/m^2: Participants were randomized to receive 60 µg/m^2 GM-CSF IV infusion. After administration of GM-CSF participant had two blisters induced on each arm followed by blood sample collection
Arm/Group | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 4
Giga cells per liter
  Session2, Day 1, 40 minutes | 0.3754 (2.78811)
  Session2, Day 1, 2 hours 40 minutes | 6.7609 (2.94642)
  Session2, Day 1, 5 hours 40 minutes | 5.8083 (1.11242)
  Session2, Day 1, 9 hours 40 minutes | 3.4558 (0.82059)
  Session2, Day 2, Pre-fluid sample | 0.4224 (1.01622)
  Session2, Day 3, Pre-fluid sample | -0.0136 (2.05134)

6. Secondary Outcome: Part 1: Change From Baseline Soluble Inflammatory Biomarkers in Skin Blister
Description: Blister samples were collected at indicated time-points for the analysis of soluble inflammatory mediators like IL-1 beta (b), Interferon-gamma (INFg), IL-6, IL-2, IL-8, Monocyte chemotactic protein-1 (MCP-1) and TNF-alpha. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. NA indicates that data was not available as standard deviation could not be calculated for a single participant.
Time Frame: Baseline; Session1: 48 hours on Day3; Session 2: 24 hours on Day 2 and 48 hours on Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Picograms per milliliter
  IL-1b, Session1, Day 3, 48 hours, n=2, 2, 2,3: number analyzed (Participants) | 2 | 2 | 2 | 3
  IL-1b, Session1, Day 3, 48 hours, n=2, 2, 2,3 | -30.9691 (3.58338) | -41.5298 (149.67553) | 3.6243 (35.28147) | 35.4452 (48.42938)
  IL-1b, Session2,Day2, 24 hours, n=2, 2, 2,1: number analyzed (Participants) | 2 | 2 | 2 | 1
  IL-1b, Session2,Day2, 24 hours, n=2, 2, 2,1 | -48.4241 (69.70779) | -83.1670 (108.13325) | 7.9733 (19.49142) | -0.3579 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  IL-1b, Session2,Day3, 48 hours, n=2, 2, 2,1: number analyzed (Participants) | 2 | 2 | 2 | 1
  IL-1b, Session2,Day3, 48 hours, n=2, 2, 2,1 | -51.0992 (46.78156) | -81.6788 (130.42664) | 7.6783 (0.42508) | -6.8302 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  IFNg, Session1,Day3, 48 hours, n=2, 0, 2, 0: number analyzed (Participants) | 2 | 0 | 2 | 0
  IFNg, Session1,Day3, 48 hours, n=2, 0, 2, 0 | 32.5244 (28.81866) |  | 55.9575 (65.86745) |
  IFNg, Session2,Day2, 24 hours, n=2, 0, 2, 0: number analyzed (Participants) | 2 | 0 | 2 | 0
  IFNg, Session2,Day2, 24 hours, n=2, 0, 2, 0 | -3.8191 (6.06240) |  | -4.5772 (7.20432) |
  IFNg, Session2,Day3, 48 hours, n=2, 0, 2, 0: number analyzed (Participants) | 2 | 0 | 2 | 0
  IFNg, Session2,Day3, 48 hours, n=2, 0, 2, 0 | 0.6652 (2.58511) |  | 2.9556 (13.15578) |
  IL-2, Session1,Day3, 48 hours, n=2, 2, 2, 3: number analyzed (Participants) | 2 | 2 | 2 | 3
  IL-2, Session1,Day3, 48 hours, n=2, 2, 2, 3 | 1.3470 (1.58747) | -0.5699 (0.80595) | 0.1623 (0.22960) | 1.2444 (1.98677)
  IL-2, Session2,Day2, 24 hours, n=2, 2, 2, 1: number analyzed (Participants) | 2 | 2 | 2 | 1
  IL-2, Session2,Day2, 24 hours, n=2, 2, 2, 1 | 0.2525 (0.66014) | 0.1804 (0.58673) | 0.0000 (0.0000) | 0.0000 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  IL-2, Session2,Day3, 48 hours, n=2, 2, 2, 1: number analyzed (Participants) | 2 | 2 | 2 | 1
  IL-2, Session2,Day3, 48 hours, n=2, 2, 2, 1 | 0.2451 (0.64975) | 2.1377 (2.64598) | 0.6968 (0.98543) | 2.1293 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  IL-6, Session1,Day3,48 hours, n=2, 0, 2, 0: number analyzed (Participants) | 2 | 0 | 2 | 0
  IL-6, Session1,Day3,48 hours, n=2, 0, 2, 0 | -1588.01 (1379.357) |  | 1535.45 (3195.182) |
  IL-6, Session2,Day2, 24 hours, n=1, 0, 1, 0: number analyzed (Participants) | 1 | 0 | 1 | 0
  IL-6, Session2,Day2, 24 hours, n=1, 0, 1, 0 | -0.13 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. |  | -349.63 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. |
  IL-6, Session2,Day3, 48 hours, n=1, 0, 2, 0: number analyzed (Participants) | 1 | 0 | 2 | 0
  IL-6, Session2,Day3, 48 hours, n=1, 0, 2, 0 | 41.39 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. |  | -25.74 (864.740) |
  IL-8, Session1,Day3,48 hours, n=2, 0, 2, 0: number analyzed (Participants) | 2 | 0 | 2 | 0
  IL-8, Session1,Day3,48 hours, n=2, 0, 2, 0 | -127550.93 (141294.871) |  | -42387.41 (31786.992) |
  IL-8, Session2,Day2, 24 hours, n=2, 0, 2, 0: number analyzed (Participants) | 2 | 0 | 2 | 0
  IL-8, Session2,Day2, 24 hours, n=2, 0, 2, 0 | -31850.03 (186366.091) |  | 34295.91 (34575.984) |
  IL-8, Session2,Day3, 48 hours, n=2, 0, 2, 0: number analyzed (Participants) | 2 | 0 | 2 | 0
  IL-8, Session2,Day3, 48 hours, n=2, 0, 2, 0 | -126387.78 (140485.270) |  | -42836.70 (30559.892) |
  MCP-1, Session1,Day3, 48 hours, n=2,4,2,4 | -36463.42 (4187.967) | -10520.93 (5858.889) | -18336.31 (9925.681) | -10284.38 (10327.369)
  MCP-1, Session2,Day2, 24 hours, n=2,4,2,4 | -2842.63 (19696.319) | 4723.83 (11253.334) | 18049.87 (1010.158) | 4299.94 (11160.896)
  MCP-1, Session2,Day3, 48 hours, n=2,4,2,4 | -18920.55 (2850.508) | 1077.95 (10014.723) | -16980.85 (11928.656) | -11416.80 (9587.163)
  TNF alpha,Session1,Day3,48 hours, n=2,2,2,3: number analyzed (Participants) | 2 | 2 | 2 | 3
  TNF alpha,Session1,Day3,48 hours, n=2,2,2,3 | -69.1140 (31.11083) | -98.8930 (55.29269) | -16.0826 (17.76133) | -33.5839 (62.80430)
  TNF alpha,Session2,Day2, 24 hours, n=2,2,2,1: number analyzed (Participants) | 2 | 2 | 2 | 1
  TNF alpha,Session2,Day2, 24 hours, n=2,2,2,1 | -25.3949 (68.42872) | 53.6996 (266.29344) | 34.8290 (63.07748) | -29.6573 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  TNF alpha,Session2,Day3,48 hours, n=2,2,2,1: number analyzed (Participants) | 2 | 2 | 2 | 1
  TNF alpha,Session2,Day3,48 hours, n=2,2,2,1 | -83.6471 (72.97148) | -110.6500 (52.29742) | -10.5091 (18.47463) | -51.9244 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant.

7. Secondary Outcome: Part 2: Change From Baseline Soluble Inflammatory Biomarkers in Skin Blister
Description: Blister samples were planned to be collected at indicated time-points for the analysis of soluble inflammatory mediators like IL-1 beta, INFg, IL-6, IL-2, IL-8, MCP-1 and TNF-alpha. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Time Frame: Baseline; Session1: 48 hours Day3; Session 2: 24 hours Day 2 and 48 hours Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Groups:
- Part 2: Participants With GM-CSF: Participants were planned to be dosed with GM-CSF (60 to a maximum dose of 480 µg/m^2) during Part 2 of the study.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Part 1: Absolute Values of Blister Volume
Description: Blister samples were collected at indicated time-points for analysis of blister volumes. . Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline.
Time Frame: Baseline, Session 1: 48 hours Day 3. Session 2: 24 hours Day 2, 48 hours Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Microliter
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Microliter
  Baseline | 361.325 (145.9115) | 156.638 (112.1876) | 185.550 (22.4860) | 230.425 (146.2442)
  Session 1, Day 3, 48 hours | 372.125 (105.8892) | 188.625 (128.1457) | 232.175 (15.0967) | 216.775 (141.8914)
  Session 2, Day 2, 24 hours | 156.225 (49.4621) | 102.838 (64.6195) | 162.975 (26.9054) | 105.363 (60.7083)
  Session 2, Day 3, 48 hours | 274.625 (110.4147) | 164.100 (104.8817) | 190.650 (10.6066) | 108.313 (79.5137)

9. Secondary Outcome: Part 2: Absolute Values of Blister Volume
Description: Blister samples were planned to be collected at indicated time-points for analysis of blister volumes. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Time Frame: Baseline, Session 1: 48 hours Day 3. Session 2: 24 hours Day 2, 48 hours Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Part 1: Change From Baseline in Cell Numbers in Blister
Description: Blister samples were collected at indicated time-points for analysis of white blood cell in blister. Latest pre-challenge LPS assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Time Frame: Baseline, Session 1: 48 hours Day 3. Session 2: 24 hours Day 2, 48 hours Day 3
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per milliliter
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg
Number analyzed (Participants) | 2 | 4 | 2
Cells per milliliter
  Session 1, Day 3, 48 hours | 841250.0 (171473.39) | -1405000.0 (6808193.03) | 667500.0 (1375322.69)
  Session 2, Day 2, 24 hours | -298750.0 (2137230.25) | -936062.5 (3258497.75) | 5447500.0 (7124100.82)
  Session 2, Day 3, 48 hours | 586250.0 (786656.29) | -1316000.0 (6556133.25) | 3275000.0 (1216223.66)

11. Secondary Outcome: Part 2: Change From Baseline in Cell Numbers in Blister
Description: Blood samples were planned to be collected at indicated time-points for analysis of white blood cell in blister. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Time Frame: Baseline, Session 1: 48 hours Day 3. Session 2: 24 hours Day 2, 48 hours Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Part 1:Change From Baseline in Cell Activation Markers by Flow Cytometry on Monocytes in Blister
Description: Blister samples were collected at indicated time-points for the measurement of activation markers by flow cytometry for monocytes in blister. Activation markers included Cluster of Differentiation (CD) 16, CD163, CD206, CD209, CD40, CD80, CD83, CD86 and Human Leukocyte Antigen - antigen D Related (HLA-DR). Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. NA indicates that data was not available as standard deviation could not be calculated for a single participant.
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Mean fluorescence intensity
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Mean fluorescence intensity
  CD16+, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 255.500 (343.6539) | 304.409 (387.9039) | 314.000 (129.4005) | 94.943 (140.1057)
  CD16+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 512.000 (515.4808) | 507.721 (375.7470) | 711.250 (942.9269) | 174.016 (226.3189)
  CD16+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 220.750 (228.0419) | -26.379 (183.4741) | 438.250 (329.1582) | 279.814 (332.5659)
  CD163+, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 1022.000 (291.3280) | 710.660 (645.7405) | 663.750 (149.5531) | 367.626 (245.5936)
  CD163+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 51.750 (217.4353) | 247.858 (249.5824) | 460.500 (120.2082) | 122.859 (88.9027)
  CD163+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 1173.750 (213.1927) | 585.093 (238.4787) | 978.750 (426.7389) | 713.995 (519.2420)
  CD206+, Session1,Day3, 48 hours, n=2, 2, 2, 4: number analyzed (Participants) | 2 | 2 | 2 | 4
  CD206+, Session1,Day3, 48 hours, n=2, 2, 2, 4 | 849.00 (3251.277) | -562.71 (207.541) | 3188.75 (5879.946) | 1295.95 (1671.924)
  CD206+, Session2,Day2, 24 hours, n=2, 0, 2, 4: number analyzed (Participants) | 2 | 0 | 2 | 4
  CD206+, Session2,Day2, 24 hours, n=2, 0, 2, 4 | 119.50 (2805.093) |  | -1224.50 (1317.340) | 9194.06 (4046.382)
  CD206+, Session2,Day3, 48 hours, n=2, 0, 2, 4: number analyzed (Participants) | 2 | 0 | 2 | 4
  CD206+, Session2,Day3, 48 hours, n=2, 0, 2, 4 | -1596.50 (823.779) |  | -1812.25 (1074.449) | 613.37 (1127.116)
  CD209+, Session1,Day3,48 hours, n=2, 4, 2, 4 | 827.000 (478.7113) | 1256.721 (676.3278) | 377.500 (457.4981) | 753.682 (482.3904)
  CD209+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 166.750 (78.8424) | 63.622 (309.3805) | 982.250 (601.3943) | 1386.776 (1523.3802)
  CD209+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 577.750 (334.8151) | 767.291 (469.9624) | 1330.250 (491.7928) | 2161.950 (1465.6418)
  CD40, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 124.750 (47.7297) | 131.238 (104.7629) | 7.500 (108.8944) | 76.408 (149.4601)
  CD40, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 200.750 (211.7785) | -60.255 (174.9309) | 116.500 (64.3467) | 436.294 (350.2183)
  CD40, Session2,Day3, 48 hours, n=1, 4, 2, 3: number analyzed (Participants) | 1 | 4 | 2 | 3
  CD40, Session2,Day3, 48 hours, n=1, 4, 2, 3 | -167.500 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant | -6.274 (238.7732) | -8.250 (42.0729) | 236.171 (304.2282)
  CD80, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 490.500 (236.1737) | 342.798 (181.3639) | 404.500 (137.8858) | 316.762 (145.7658)
  CD80, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 155.250 (284.6105) | 50.962 (31.2323) | 44.250 (158.0384) | 44.488 (94.3934)
  CD80, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 286.250 (14.4957) | 324.662 (223.8334) | 254.000 (77.7817) | 401.521 (43.5362)
  CD83, Session1,Day3, 48 hours, n=2, 4, 2, 4 | -832.500 (89.8026) | -816.619 (242.1554) | -373.250 (578.7669) | -824.574 (521.9010)
  CD83, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 83.250 (361.6851) | 44.949 (222.8885) | 791.500 (1207.0313) | 280.947 (870.1350)
  CD83, Session2,Day3, 48 hours, n=2, 4, 2, 4 | -978.250 (339.0577) | -773.455 (383.3063) | -328.250 (171.4734) | -529.900 (854.9675)
  CD86+, Session1,Day3, 48 hours, n=2, 4, 2, 4 | -439.750 (195.5150) | -51.662 (369.1392) | -319.750 (71.7713) | -497.468 (327.7072)
  CD86+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | -275.500 (30.4056) | -241.591 (286.2295) | 103.750 (15.9099) | 6.398 (418.6691)
  CD86+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | -723.250 (104.2983) | 312.288 (458.1399) | -292.250 (16.6170) | -97.004 (1081.7203)
  HLA-DR, Session1,Day3, 48 hours, n=2, 4, 2, 4 | -5189.00 (2028.689) | -3291.05 (4596.102) | -7267.75 (11655.595) | -2543.35 (3800.276)
  HLA-DR, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 388.50 (3168.545) | -9344.96 (2661.368) | -2229.25 (4812.922) | 10097.91 (12898.982)
  HLA-DR, Session2,Day3, 48 hours, n=2, 4, 2, 4 | -7846.25 (6101.978) | -10329.79 (4408.080) | -9340.00 (10061.422) | 8884.70 (15377.757)

13. Secondary Outcome: Part 2:Change From Baseline in Cell Activation Markers by Flow Cytometry on Monocytes in Blister
Description: Blister samples were planned to be collected at indicated time-points for the measurement of activation. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Part 1:Change From Baseline of CD40+/CD80+ by Flow Cytometry on Monocytes in Blister
Description: Blister samples were collected at indicated time-points for the measurement of activation markers by flow cytometry for monocytes in blister like CD40+/CD80+. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. NA indicates that data was not available as standard deviation could not be calculated for a single participant.
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Ratio
  Session1,Day3, 48 hours, n=2, 4, 2, 4 | 0.1475 (0.22981) | 0.2764 (0.19587) | 0.0610 (0.13294) | -0.4060 (0.82999)
  Session2,Day2, 24 hours, n=2, 4, 2, 4 | 0.0925 (0.15203) | 0.5062 (0.70807) | 0.5108 (0.67069) | -0.0994 (1.34749)
  Session2,Day3, 48 hours, n=1, 4, 2, 3: number analyzed (Participants) | 1 | 4 | 2 | 3
  Session2,Day3, 48 hours, n=1, 4, 2, 3 | -0.1210 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | 0.3015 (0.39252) | 0.1300 (0.03748) | -0.2698 (1.09270)

15. Secondary Outcome: Part 2:Change From Baseline of CD40+/CD80+ by Flow Cytometry on Monocytes in Blister
Description: as for outcome 13
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Part 1:Change From Baseline in Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blister
Description: Blister samples were collected at indicated time-points for the measurement of activation markers by flow cytometry for dendritic cells in blister. Activation markers included CD16, CD163, CD206, CD209, CD40, CD80, CD83, CD86 and HLA-DR. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. NA indicates that data was not available as standard deviation could not be calculated for a single participant.
Time Frame: Baseline; Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Mean fluorescence intensity
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Mean fluorescence intensity
  CD16+, Session1,Day3, 48 hours, n=2, 4, 2, 4 | -31.250 (48.4368) | 668.512 (634.0204) | 44.500 (90.5097) | 83.647 (119.1684)
  CD16+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 284.750 (2.4749) | 235.293 (200.9269) | 62.750 (48.4368) | 225.589 (233.9677)
  CD16+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 154.000 (44.5477) | 208.225 (339.7035) | 186.250 (254.9120) | 268.838 (315.3551)
  CD163+, Session1,Day3, 48 hours, n=2, 4, 2, 4 | -103.7500 (129.04699) | -91.1420 (123.34114) | -105.7500 (107.83378) | -16.6220 (31.79210)
  CD163+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | -112.7500 (143.89623) | -49.4854 (72.90224) | 267.2500 (66.11448) | 47.1343 (60.71649)
  CD163+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | -132.2500 (119.85460) | -124.5144 (79.57686) | -70.0000 (101.11627) | -32.4464 (30.09999)
  CD206+, Session1,Day3, 48 hours, n=2, 2, 2, 4: number analyzed (Participants) | 2 | 2 | 2 | 4
  CD206+, Session1,Day3, 48 hours, n=2, 2, 2, 4 | -56.00 (601.041) | -1057.04 (1641.526) | 1372.75 (2325.321) | 2032.27 (1708.909)
  CD206+, Session2,Day2, 24 hours, n=2, 0, 2, 4: number analyzed (Participants) | 2 | 0 | 2 | 4
  CD206+, Session2,Day2, 24 hours, n=2, 0, 2, 4 | -430.25 (1407.496) |  | -665.00 (481.540) | 3032.02 (3183.213)
  CD206+, Session2,Day3, 48 hours, n=2, 0, 2, 4: number analyzed (Participants) | 2 | 0 | 2 | 4
  CD206+, Session2,Day3, 48 hours, n=2, 0, 2, 4 | 4.00 (171.120) |  | 198.75 (150.260) | 856.32 (1654.671)
  CD209+, Session1,Day3,48 hours, n=2, 4, 2, 4 | 83.250 (15.2028) | 765.140 (690.4086) | -211.000 (17.6777) | 95.101 (191.7562)
  CD209+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 79.750 (37.1231) | 38.604 (582.9139) | 743.750 (482.6004) | 1834.867 (1573.3002)
  CD209+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 101.750 (341.1790) | 297.936 (605.5896) | 835.000 (444.7702) | 1822.510 (1522.9886)
  CD40, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 963.750 (110.6622) | 1403.000 (754.2476) | 776.000 (30.4056) | 923.024 (560.8252)
  CD40, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 96.000 (266.5793) | 17.354 (257.3845) | -10.250 (61.1647) | 293.485 (249.0144)
  CD40, Session2,Day3, 48 hours, n=1, 4, 2, 3: number analyzed (Participants) | 1 | 4 | 2 | 3
  CD40, Session2,Day3, 48 hours, n=1, 4, 2, 3 | 383.500 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | 1072.416 (523.9965) | 783.750 (127.6328) | 1389.536 (710.1286)
  CD80, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 2609.000 (376.8879) | 4155.674 (893.4273) | 2366.000 (72.8320) | 4998.865 (1326.4663)
  CD80, Session2,Day2, 24 hours, n=2, 4, 2, 4 | -130.000 (523.2590) | -583.016 (1305.3774) | -237.250 (252.0836) | 407.277 (615.0693)
  CD80, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 1235.000 (603.8692) | 3665.666 (1565.6126) | 1407.250 (331.9866) | 3958.838 (803.7564)
  CD83, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 2342.250 (423.2034) | 2806.835 (741.9070) | 2624.000 (770.7464) | 3834.100 (1511.6374)
  CD83, Session2,Day2, 24 hours, n=2, 4, 2, 4 | -28.000 (656.9022) | -409.187 (1498.2826) | -343.250 (597.1517) | 648.346 (685.4282)
  CD83, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 1199.500 (900.8540) | 3368.105 (953.2468) | 2924.250 (510.1775) | 3264.300 (988.2407)
  CD86+, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 2590.75 (1485.278) | 4689.54 (1189.323) | 2701.50 (65.761) | 3936.29 (2537.066)
  CD86+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | -509.75 (345.422) | -696.70 (1551.690) | -184.00 (373.352) | 94.29 (782.682)
  CD86+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 1175.25 (980.404) | 7229.67 (2733.004) | 2750.50 (421.436) | 4132.68 (2423.146)
  HLA-DR, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 1020.00 (2766.909) | 31657.05 (11524.385) | -2661.75 (19339.017) | 3242.86 (11323.629)
  HLA-DR, Session2,Day2, 24 hours, n=2, 4, 2, 4 | -494.00 (1211.981) | -3470.23 (16869.569) | 480.50 (11477.050) | 11902.82 (17969.677)
  HLA-DR, Session2,Day3, 48 hours, n=2, 4, 2, 4 | -4386.50 (911.461) | 16282.97 (22938.047) | 1564.00 (12854.494) | 19351.27 (16136.948)

17. Secondary Outcome: Part 2:Change From Baseline in Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blister
Description: as for outcome 13
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Part 1:Change From Baseline of CD40+/CD80+ by Flow Cytometry on Dendritic Cells in Blister
Description: Blister samples were collected at indicated time-points for the measurement of activation markers by flow cytometry for dendritic cells in blister like CD40+/CD80+. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. NA indicates that data was not available as standard deviation could not be calculated for a single participant.
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Ratio
  Session1,Day3, 48 hours, n=2, 4, 2, 4 | 42.7675 (5.32805) | 43.2094 (6.81783) | 47.8100 (4.17193) | 39.8453 (6.60325)
  Session2,Day2, 24 hours, n=2, 4, 2, 4 | 2.7250 (14.65125) | 0.0825 (18.06488) | 0.0900 (1.52735) | 6.7523 (9.76233)
  Session2,Day3, 48 hours, n=1, 4, 2, 3: number analyzed (Participants) | 1 | 4 | 2 | 3
  Session2,Day3, 48 hours, n=1, 4, 2, 3 | 27.7000 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | 42.6493 (11.60035) | 42.5100 (2.82843) | 38.4313 (6.81975)

19. Secondary Outcome: Part 2:Change From Baseline of CD40+/CD80+ by Flow Cytometry on Dendritic Cells in Blister
Description: as for outcome 13
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Part 1:Change From Baseline in Cell Activation Markers by Flow Cytometry on Macrophages in Blister
Description: Blister samples were collected at indicated time-points for the measurement of activation markers by flow cytometry for macrophages in blister. Activation markers included CD16, CD163, CD206, CD209, CD40, CD80, CD83, CD86 and HLA-DR. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. NA indicates that data was not available as standard deviation could not be calculated for a single participant.
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Mean fluorescence intensity
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Mean fluorescence intensity
  CD16+, Session1,Day3, 48 hours, n=2, 4, 2, 4 | -5027.00 (5289.866) | 4510.75 (7162.125) | -3449.75 (1895.400) | -2607.25 (6559.210)
  CD16+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 13111.25 (32672.929) | -2948.25 (3659.787) | 5372.75 (235.113) | -1010.00 (5492.201)
  CD16+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | -4621.75 (8382.397) | -6203.50 (13105.657) | -3286.25 (947.170) | -3653.63 (5345.655)
  CD163+, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 888.500 (292.0351) | 400.500 (455.9359) | 270.250 (97.9343) | 723.125 (717.7969)
  CD163+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 49.750 (215.3140) | 48.250 (163.7506) | 415.250 (142.4820) | 169.750 (160.7060)
  CD163+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 1012.000 (501.3387) | 411.000 (524.8443) | 719.250 (63.9932) | 789.513 (825.7539)
  CD206+, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 81.00 (2206.173) | -1275.50 (3073.903) | -955.75 (1183.343) | -734.88 (5799.935)
  CD206+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 4503.00 (9540.992) | 564.00 (2911.625) | -1329.50 (1668.065) | 12596.63 (16264.004)
  CD206+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | -1229.25 (973.332) | -2542.63 (4084.922) | -2193.50 (543.765) | -2622.75 (3423.992)
  CD209+, Session1,Day3,48 hours, n=2, 4, 2, 4 | 931.00 (505.581) | 458.88 (1827.032) | -333.00 (416.486) | 890.88 (2206.644)
  CD209+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 474.75 (485.429) | 21.63 (1282.820) | 1672.25 (1038.386) | 5641.13 (4969.374)
  CD209+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 565.75 (840.396) | -236.13 (1413.395) | 1607.75 (1283.752) | 2835.13 (2917.207)
  CD40, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 593.25 (20.860) | 198.00 (1021.994) | 371.75 (1282.338) | -59.50 (536.615)
  CD40, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 1007.00 (1119.350) | -43.38 (837.351) | -691.50 (542.351) | 3426.13 (4547.393)
  CD40, Session2,Day3, 48 hours, n=1, 4, 2, 4: number analyzed (Participants) | 1 | 4 | 2 | 4
  CD40, Session2,Day3, 48 hours, n=1, 4, 2, 4 | 74.50 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | -166.13 (503.207) | -480.25 (925.956) | -70.50 (1739.426)
  CD80, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 884.00 (9.899) | 1193.63 (1486.267) | 1403.75 (3760.040) | 304.88 (2126.019)
  CD80, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 1250.50 (1339.967) | 353.63 (2446.460) | -1136.25 (1490.935) | 1215.88 (2013.518)
  CD80, Session2,Day3, 48 hours, n=2, 4, 2, 4 | -84.75 (23.688) | -114.50 (615.327) | -1686.50 (2957.121) | -744.88 (3479.863)
  CD83, Session1,Day3, 48 hours, n=2, 4, 2, 4 | -1139.00 (477.297) | -556.88 (1063.877) | 2522.00 (1359.766) | -842.63 (1505.636)
  CD83, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 420.50 (3235.014) | 1243.25 (3307.491) | 2690.50 (4319.008) | 918.75 (1945.597)
  CD83, Session2,Day3, 48 hours, n=2, 4, 2, 4 | -1703.75 (15.203) | -1046.38 (561.034) | 745.75 (496.743) | -1668.63 (2068.363)
  CD86+, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 792.50 (338.704) | 577.50 (1141.719) | 2311.50 (1262.186) | 28.25 (2057.408)
  CD86+, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 381.25 (2896.663) | 674.50 (1496.032) | -329.75 (197.636) | -570.75 (3118.314)
  CD86+, Session2,Day3, 48 hours, n=2, 4, 2, 4 | 13.75 (285.318) | 1692.50 (1687.192) | 181.75 (506.642) | 517.50 (5171.981)
  HLA-DR, Session1,Day3, 48 hours, n=2, 4, 2, 4 | 3326.25 (1854.388) | -7695.38 (19317.582) | 6003.75 (17276.386) | -5724.25 (49407.676)
  HLA-DR, Session2,Day2, 24 hours, n=2, 4, 2, 4 | 7435.25 (35884.608) | 13061.88 (29527.416) | 1273.75 (3391.638) | 36041.13 (33139.756)
  HLA-DR, Session2,Day3, 48 hours, n=2, 4, 2, 4 | -882.00 (1575.434) | -20377.25 (25175.815) | -8397.75 (19009.505) | 11460.13 (56951.939)

21. Secondary Outcome: Part 2:Change From Baseline in Cell Activation Markers by Flow Cytometry on Macrophages in Blister
Description: as for outcome 13
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Part 1:Change From Baseline of CD40+/CD80+ by Flow Cytometry on Macrophages in Blister
Description: as for outcome 18
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Ratio
  Session1,Day3, 48 hours, n=2, 4, 2, 4 | 11.0475 (9.89596) | -1.2837 (17.00275) | 21.8500 (26.44579) | -0.8938 (20.18664)
  Session2,Day2, 24 hours, n=2, 4, 2, 4 | 15.1225 (35.88213) | 1.3537 (22.85581) | -16.0250 (3.35876) | 9.1137 (15.78332)
  Session2,Day3, 48 hours, n=1, 4, 2, 4: number analyzed (Participants) | 1 | 4 | 2 | 4
  Session2,Day3, 48 hours, n=1, 4, 2, 4 | 0.3500 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | -2.9838 (10.58741) | -8.9750 (17.00592) | -3.2238 (27.65006)

23. Secondary Outcome: Part 2:Change From Baseline of CD40+/CD80+ by Flow Cytometry on Macrophages in Blister
Description: as for outcome 13
Time Frame: Baseline, Session1: 48 hours Day 3, Session 2: 24 hours Day 2 and 48 hours Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Part 1:Change From Baseline in Soluble Inflammatory Mediators in Blood
Description: Blood samples were collected at indicated timepoints for the analysis of primary soluble inflammatory mediators like IL-1 beta, INFg, IL-2, IL-8, and MCP-1 in blood. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. NA indicates that data was not available as standard deviation could not be calculated for a single participant.
Time Frame: Baseline, Session 2: -5, 10, 25, 40 minutes, 1 hour 10 minutes, 1 hour 40 minutes, 2 hours 40 minutes, 5 hours 40 minutes on Day 1. Pre-fluid sample on Day 2 and Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Picograms per milliliter
  INFg, Session2,Day1, -5 minutes, n=2, 4, 2, 4 | -0.5636 (0.24961) | -0.1278 (0.23076) | 0.0653 (0.80201) | 5.7255 (1.85029)
  INFg, Session2,Day1, 10 minutes, n=2, 4, 2, 4 | -0.4140 (0.05250) | -0.3298 (0.20362) | -0.2355 (0.28729) | 6.0071 (1.26842)
  INFg, Session2,Day1, 25 minutes, n=1, 4, 2, 4: number analyzed (Participants) | 1 | 4 | 2 | 4
  INFg, Session2,Day1, 25 minutes, n=1, 4, 2, 4 | -0.6996 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | -0.3697 (0.19518) | -0.2432 (0.30593) | 6.1605 (1.77144)
  INFg, Session2,Day1, 40 minutes, n=2, 4, 2, 4 | -0.6745 (0.26829) | -0.4771 (0.41990) | 0.1501 (0.28816) | 5.4142 (2.07138)
  INFg, Session2,Day1, 1 hour 10 minutes, n=2, 4,2,4 | 1.8597 (2.47610) | 1.7673 (1.80932) | 6.6083 (0.78111) | 4.9508 (1.77082)
  INFg, Session2,Day1, 1 hour 40 minutes, n=2, 4,2,4 | 6.5709 (5.72091) | 6.5863 (3.69982) | 13.6809 (3.56564) | 3.8804 (2.00819)
  INFg, Session2,Day1, 2 hour 40 minutes, n=2, 4,2,4 | 9.1319 (7.94104) | 8.7498 (2.97730) | 15.7306 (3.51048) | 2.7181 (2.63053)
  INFg, Session2,Day1, 5 hour 40 minutes, n=2, 4,2,4 | 3.5927 (3.83382) | 3.2672 (1.86587) | 5.0294 (3.92184) | 1.7041 (1.64895)
  INFg, Session2,Day2, Pre-fluid sampling, n=2,4,2,4 | -3.7611 (1.04373) | 0.7630 (1.43167) | -0.3514 (1.05828) | -3.0755 (2.76516)
  INFg, Session2,Day3, Pre-fluid sampling, n=2,4,2,4 | -4.3628 (0.31014) | 1.5962 (3.09933) | -2.6600 (1.75306) | -3.2817 (2.72811)
  IL-1b, Session2,Day1, -5 minutes, n=2, 4, 2,4 | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000)
  IL-1b, Session2,Day1, 10 minutes, n=2, 4, 2,4 | 0.0000 (0.0000) | 0.0008 (0.00150) | 0.0000 (0.0000) | 0.0000 (0.0000)
  IL-1b, Session2,Day1, 25 minutes, n=1, 4, 2,4: number analyzed (Participants) | 1 | 4 | 2 | 4
  IL-1b, Session2,Day1, 25 minutes, n=1, 4, 2,4 | 0.0000 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | 0.0000 (0.00000) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-1b, Session2,Day1, 40 minutes, n=2, 4, 2,4 | 0.0000 (0.00000) | 0.0008 (0.00150) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-1b, Session2,Day1, 1hour 10minutes, n=2,4,2,4 | 0.0000 (0.00000) | 0.0008 (0.00150) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-1b, Session2,Day1, 1hour 40minutes, n=2,4,2,4 | 0.0000 (0.00000) | 0.1875 (0.37303) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-1b, Session2,Day1, 2hour 40minutes, n=2,4,2,4 | 0.0000 (0.00000) | 0.3194 (0.41468) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-1b, Session2,Day1, 5hour 40minutes, n=2,4,2,4 | 0.0000 (0.00000) | 0.0008 (0.00150) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-1b, Session2,Day2,Pre-fluid sample, n=2,4,2,4 | 0.2225 (0.31897) | 0.0008 (0.00150) | -0.0030 (0.00000) | 0.0857 (0.10517)
  IL-1b, Session2,Day3,Pre-fluid sample, n=2,4,2,4 | -0.0030 (0.00000) | 0.0008 (0.00150) | -0.0030 (0.00000) | -0.0015 (0.00173)
  IL-2, Session2,Day1, -5 minutes, n=0, 4, 2,4: number analyzed (Participants) | 0 | 4 | 2 | 4
  IL-2, Session2,Day1, -5 minutes, n=0, 4, 2,4 |  | 0.0000 (0.00000) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-2, Session2,Day1, 10 minutes, n=0, 4, 2,2: number analyzed (Participants) | 0 | 4 | 2 | 2
  IL-2, Session2,Day1, 10 minutes, n=0, 4, 2,2 |  | 0.0031 (0.00625) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-2, Session2,Day1, 25 minutes, n=0, 4, 2,4: number analyzed (Participants) | 0 | 4 | 2 | 4
  IL-2, Session2,Day1, 25 minutes, n=0, 4, 2,4 |  | 0.0031 (0.00625) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-2, Session2,Day1, 40 minutes, n=0, 3, 2,2: number analyzed (Participants) | 0 | 3 | 2 | 2
  IL-2, Session2,Day1, 40 minutes, n=0, 3, 2,2 |  | 0.0000 (0.00000) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-2, Session2,Day1, 1 hour 10 minutes, n=0, 4,2,4: number analyzed (Participants) | 0 | 4 | 2 | 4
  IL-2, Session2,Day1, 1 hour 10 minutes, n=0, 4,2,4 |  | 0.0031 (0.00625) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-2, Session2,Day1, 1 hour 40 minutes, n=0, 4,2,2: number analyzed (Participants) | 0 | 4 | 2 | 2
  IL-2, Session2,Day1, 1 hour 40 minutes, n=0, 4,2,2 |  | 0.0031 (0.00625) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-2, Session2,Day1, 2 hour 40 minutes, n=0, 4,2,2: number analyzed (Participants) | 0 | 4 | 2 | 2
  IL-2, Session2,Day1, 2 hour 40 minutes, n=0, 4,2,2 |  | 0.0031 (0.00625) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-2, Session2,Day1, 5 hour 40 minutes, n=0, 4,2,2: number analyzed (Participants) | 0 | 4 | 2 | 2
  IL-2, Session2,Day1, 5 hour 40 minutes, n=0, 4,2,2 |  | 0.0031 (0.00625) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IL-2, Session2,Day2, Pre-fluid sampling, n=2,4,2,4 | 0.0000 (0.00000) | 0.0031 (0.00625) | -0.0160 (0.00000) | -0.0018 (0.01645)
  IL-2, Session2,Day3, Pre-fluid sampling, n=2,4,2,4 | 0.0000 (0.00000) | 0.0031 (0.00625) | -0.0160 (0.00000) | -0.0018 (0.01645)
  IL-8, Session2,Day1, -5 minutes, n=2, 4, 2,4 | -1.4835 (2.97824) | 0.0761 (0.99505) | 0.1849 (0.08020) | 83.1531 (44.11662)
  IL-8, Session2,Day1, 10 minutes, n=2, 4, 2,4 | 2.2890 (3.42770) | 0.0714 (1.30027) | 0.8613 (0.83194) | 89.0123 (48.41011)
  IL-8, Session2,Day1, 25 minutes, n=1, 4, 2,4: number analyzed (Participants) | 1 | 4 | 2 | 4
  IL-8, Session2,Day1, 25 minutes, n=1, 4, 2,4 | 1.7998 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | 0.6814 (1.27650) | 3.0142 (1.22739) | 86.4178 (47.57975)
  IL-8, Session2,Day1, 40 minutes, n=2, 3, 2,4: number analyzed (Participants) | 2 | 3 | 2 | 4
  IL-8, Session2,Day1, 40 minutes, n=2, 3, 2,4 | 9.4905 (1.93306) | 9.3036 (5.86829) | 27.1507 (3.96686) | 50.4514 (20.49601)
  IL-8, Session2,Day1, 1 hour 10 minutes, n=2, 3,2,4: number analyzed (Participants) | 2 | 3 | 2 | 4
  IL-8, Session2,Day1, 1 hour 10 minutes, n=2, 3,2,4 | 105.0587 (43.02522) | 141.7558 (104.21164) | 162.3033 (42.93991) | 76.6709 (36.79748)
  IL-8, Session2,Day1, 1 hour 40 minutes, n=2,3, 2,4: number analyzed (Participants) | 2 | 3 | 2 | 4
  IL-8, Session2,Day1, 1 hour 40 minutes, n=2,3, 2,4 | 214.1372 (181.31639) | 468.8635 (296.06234) | 229.6116 (155.88116) | 77.3493 (73.83422)
  IL-8, Session2,Day1, 2 hour 40 minutes, n=2,3, 2,4: number analyzed (Participants) | 2 | 3 | 2 | 4
  IL-8, Session2,Day1, 2 hour 40 minutes, n=2,3, 2,4 | 49.6247 (26.76026) | 340.0657 (234.74182) | 111.6155 (118.63027) | 126.3552 (204.81735)
  IL-8, Session2,Day1, 5 hour 40 minutes, n=2,3, 2,4: number analyzed (Participants) | 2 | 3 | 2 | 4
  IL-8, Session2,Day1, 5 hour 40 minutes, n=2,3, 2,4 | 7.6772 (3.55867) | 88.5574 (24.09240) | 19.5090 (6.86764) | 30.1483 (10.71198)
  IL-8, Session2,Day2, Pre-fluid sampling, n=2,3,2,4: number analyzed (Participants) | 2 | 3 | 2 | 4
  IL-8, Session2,Day2, Pre-fluid sampling, n=2,3,2,4 | 3.8330 (7.21699) | 8.7544 (16.57327) | -1.3116 (1.93618) | 33.5296 (54.13468)
  IL-8, Session2,Day3, Pre-fluid sampling, n=2,4,2,4 | -1.3819 (2.32148) | 0.6465 (2.78896) | -0.8507 (0.69264) | -2.0468 (1.21979)
  MCP-1, Session2,Day1, -5 minutes, n=2, 4, 2,4 | -1.984 (0.9353) | 7.280 (11.0662) | -12.078 (6.4316) | 2702.736 (1675.5428)
  MCP-1, Session2,Day1, 10 minutes, n=2, 4, 2,4 | 1.716 (33.8987) | 15.335 (18.3588) | -6.963 (11.3479) | 3692.647 (1671.9037)
  MCP-1, Session2,Day1, 25 minutes, n=1, 4, 2,4: number analyzed (Participants) | 1 | 4 | 2 | 4
  MCP-1, Session2,Day1, 25 minutes, n=1, 4, 2,4 | -25.166 (NA) — NA indicates that data was not available as standard deviation could not be calculated for a single participant. | 22.679 (14.0540) | 9.360 (10.2709) | 4354.050 (1579.4757)
  MCP-1, Session2,Day1, 40 minutes, n=2, 4, 2,4 | 53.774 (44.7737) | 108.005 (54.2180) | 273.261 (29.0646) | 4218.511 (1850.5204)
  MCP-1, Session2,Day1, 1 hour 10 minutes, n=2,4,2,4 | 1092.558 (576.0879) | 3281.560 (2188.7631) | 2993.718 (17.3345) | 4119.865 (2047.7930)
  MCP-1, Session2,Day1, 1 hour 40 minutes, n=2,4,2,4 | 2521.255 (1886.7927) | 5164.946 (25.3073) | 6182.663 (13.9688) | 2659.013 (1778.3867)
  MCP-1, Session2,Day1, 2 hour 40 minutes, n=2,4,2,4 | 1449.223 (880.4065) | 5189.946 (75.0973) | 6824.798 (3014.6330) | 1405.284 (603.0458)
  MCP-1, Session2,Day1, 5 hour 40 minutes, n=2,4,2,4 | 126.224 (72.8644) | 588.424 (384.1274) | 350.071 (81.7289) | 365.641 (156.6637)
  MCP-1, Session2,Day2,Pre-fluid sampling, n=2,4,2,4 | -0.963 (23.0612) | 38.016 (54.7584) | -2.917 (42.8500) | -14.427 (32.7430)
  MCP-1, Session2,Day3,Pre-fluid sampling, n=2,4,2,4 | -12.333 (0.9485) | 28.822 (23.2955) | 8.210 (9.0286) | -15.571 (25.0756)

25. Secondary Outcome: Part 2:Change From Baseline in Soluble Inflammatory Mediators in Blood
Description: Blood samples were planned to be collected at indicated time-points for the measurement of activation. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Time Frame: as for outcome 24
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Part 1: Change From Baseline in Soluble Inflammatory Mediators in Blood: TNF-alpha, IL-6 and GM-CSF: GM-CSF Arm
Description: Blood samples were collected at indicated time-points for the analysis of soluble inflammatory mediators like TNF-alpha, IL-6 and GM-CSF in blood. Latest pre-challenge GM-CSF assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Time Frame: as for outcome 24
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 4
Picograms per milliliter
  GM-CSF, Session2,Day1, -5 minutes | 1674.235 (635.9050)
  GM-CSF, Session2,Day1, 10 minutes | 1260.988 (850.1777)
  GM-CSF, Session2,Day1, 25 minutes: number analyzed (Participants) | 1
  GM-CSF, Session2,Day1, 25 minutes | 624.895 (287.0075)
  GM-CSF, Session2,Day1, 40 minutes | 364.045 (218.4348)
  GM-CSF, Session2,Day1,1 hour 10 minutes | 145.793 (97.7248)
  GM-CSF, Session2,Day1,1 hour 40 minutes | 52.158 (39.5878)
  GM-CSF, Session2,Day1,2 hour 40 minutes | 7.486 (9.9232)
  GM-CSF, Session2,Day1,5 hour 40 minutes | 0.000 (0.0000)
  GM-CSF, Session2,Day2,Pre-fluid sampling | 0.000 (0.0000)
  GM-CSF, Session2,Day3,Pre-fluid sampling | 0.000 (0.0000)
  IL-6, Session2,Day1, -5 minutes | 8.8136 (3.54771)
  IL-6, Session2,Day1, 10 minutes | 11.3851 (1.98376)
  IL-6, Session2,Day1, 25 minutes | 13.0699 (3.47569)
  IL-6, Session2,Day1, 40 minutes | 10.9359 (5.03738)
  IL-6, Session2,Day1, 1hour 10minutes | 6.8485 (3.17943)
  IL-6, Session2,Day1, 1hour 40minutes | 5.0334 (2.72854)
  IL-6, Session2,Day1, 2hour 40minutes | 2.6496 (1.56258)
  IL-6, Session2,Day1, 5hour 40minutes | 1.9135 (1.60586)
  IL-6, Session2,Day2,Pre-fluid sample | 1.2598 (1.72396)
  IL-6, Session2,Day3,Pre-fluid sample | -0.0324 (0.13824)
  TNF-alpha, Session2,Day1, -5 minutes | 2.6740 (0.39814)
  TNF-alpha, Session2,Day1, 10 minutes | 2.4860 (0.70400)
  TNF-alpha, Session2,Day1, 25 minutes | 2.5475 (0.86898)
  TNF-alpha, Session2,Day1, 40 minutes | 2.2100 (0.99729)
  TNF-alpha, Session2,Day1, 1 hour 10 minutes | 2.1380 (0.90651)
  TNF-alpha, Session2,Day1, 1 hour 40 minutes | 1.9665 (1.19555)
  TNF-alpha, Session2,Day1, 2 hour 40 minutes | 1.6001 (0.80929)
  TNF-alpha, Session2,Day1, 5 hour 40 minutes | 0.9562 (0.63271)
  TNF-alpha, Session2,Day2, Pre-fluid sampling | 0.5423 (0.50847)
  TNF-alpha, Session2,Day3, Pre-fluid sampling | -0.1194 (0.55216)

27. Secondary Outcome: Part 2: Change From Baseline in Soluble Inflammatory Mediators in Blood: TNF-alpha, IL-6 and GM-CSF for GM-CSF Arm
Description: Blood samples were planned to be collected at indicated time-points for the measurement of activation. Latest pre-challenge GM-CSF assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Time Frame: as for outcome 24
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0

28. Secondary Outcome: Part 1: Change From Baseline in Soluble Inflammatory Mediators in Blood: C-reactive Protein (CRP)
Description: Blood samples were collected at indicated time-points for the analysis of soluble inflammatory mediators like CRP in blood. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Time Frame: Baseline; Session 2: Post challenge Day 1. Pre-fluid sample on Day 2 and Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Milligrams per liter
  Session2,Day1, Post-challenge | 0.20 (3.111) | 2.75 (0.624) | 2.40 (0.990) | 1.53 (0.457)
  Session2,Day 2, Pre-fluid sample | 7.50 (4.667) | 21.80 (2.380) | 18.55 (4.455) | 5.80 (1.623)
  Session2,Day 3, Pre-fluid sample | 1.50 (3.111) | 10.65 (0.968) | 8.45 (0.636) | 2.25 (0.451)

29. Secondary Outcome: Part 2: Change From Baseline in Soluble Inflammatory Mediators in Blood: CRP
Description: as for outcome 25
Time Frame: Baseline; Session 2: Post challenge Day 1; Pre-fluid sample on Day 2 and Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Part 1: Change From Baseline in Cell Activation Markers by Flow Cytometry on Monocytes in Blood
Description: Blood samples were collected at indicated time-points for the measurement of activation markers by flow cytometry for monocytes in blood. Activation markers included CD16, CD163, CD206, CD209, CD40, CD80, CD83, CD86 and HLA-DR. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Time Frame: Baseline; Session 2: 40 minutes, 2 hours 40 minutes, 5 hours 40 minutes, 9 hours 40 minutes on Day 1. Pre-fluid sample on Day 2 and Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Mean fluorescence intensity
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Mean fluorescence intensity
  CD16+, Session2,Day1, 40 minutes, n=2, 4, 2,4 | -117.5000 (55.86144) | -10.5565 (50.64061) | -47.0000 (39.59798) | -26.3505 (10.83082)
  CD16+, Session2,Day1, 2 hour 40 minutes, n=2,4,2,4 | -128.9500 (131.45115) | -31.4965 (41.99141) | -76.6000 (69.29646) | -26.6015 (13.40656)
  CD16+, Session2,Day1, 5 hour 40 minutes, n=2,4,2,4 | -130.1500 (78.98383) | -35.3433 (40.19923) | -94.3000 (56.85139) | -29.1195 (15.07448)
  CD16+, Session2,Day1,9 hour 40 minutes,n-0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD16+, Session2,Day1,9 hour 40 minutes,n-0,0,0,4 |  |  |  | -24.5510 (13.98978)
  CD16+,Session2,Day2, Pre-fluid sampling, n=2,4,2,4 | 125.5000 (47.37615) | 162.8120 (171.51836) | 427.5000 (132.22897) | 42.9945 (58.62985)
  CD16+,Session2,Day3, Pre-fluid sampling, n=2,4,2,4 | -24.5000 (40.30509) | -6.6285 (33.04476) | 142.5000 (71.41778) | -11.7065 (24.07118)
  CD163+, Session2,Day1, 40 minutes, n=2,4,2,4 | -371.000 (199.4041) | -833.203 (131.9463) | -721.000 (131.5219) | -511.618 (152.8883)
  CD163+, Session2,Day1,2 hour 40 minutes, n=2,4,2,4 | -499.500 (147.7853) | -902.203 (205.5423) | -790.000 (8.4853) | -426.253 (144.1939)
  CD163+, Session2,Day1,5 hour 40 minutes, n=2,4,2,4 | -363.500 (112.4300) | -694.390 (222.5211) | -522.500 (112.4300) | -376.659 (156.2613)
  CD163+, Session2,Day1, 9 hour 40 minutes,n-0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD163+, Session2,Day1, 9 hour 40 minutes,n-0,0,0,4 |  |  |  | -314.464 (132.3300)
  CD163+,Session2,Day2, Pre-fluid sampling,n=2,4,2,4 | 4.500 (19.0919) | 146.403 (737.3912) | 22.500 (225.5671) | -73.247 (127.0624)
  CD163+,Session2,Day3, Pre-fluid sampling,n=2,4,2,4 | -66.000 (8.4853) | 3.801 (244.5535) | -80.000 (66.4680) | 63.254 (54.8309)
  CD206+, Session2,Day1, 40 minutes, n=2,3,2,4: number analyzed (Participants) | 2 | 3 | 2 | 4
  CD206+, Session2,Day1, 40 minutes, n=2,3,2,4 | -502.500 (171.8269) | -892.543 (205.7220) | 86.500 (263.7508) | 932.807 (829.8233)
  CD206+, Session2,Day1,2 hour 40 minutes, n=2,2,2,4: number analyzed (Participants) | 2 | 2 | 2 | 4
  CD206+, Session2,Day1,2 hour 40 minutes, n=2,2,2,4 | 1011.000 (2743.5743) | -583.485 (672.1029) | -293.500 (102.5305) | 1808.345 (1763.3758)
  CD206+, Session2,Day1,5 hour 40 minutes, n=2,2,2,4: number analyzed (Participants) | 2 | 2 | 2 | 4
  CD206+, Session2,Day1,5 hour 40 minutes, n=2,2,2,4 | -388.500 (74.2462) | -686.465 (521.9367) | 12.000 (309.7128) | 2051.872 (858.1801)
  CD206+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD206+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | 2546.884 (2810.2028)
  CD206+,Session2,Day2, Pre-fluid sampling,n=2,2,2,4: number analyzed (Participants) | 2 | 2 | 2 | 4
  CD206+,Session2,Day2, Pre-fluid sampling,n=2,2,2,4 | 423.000 (196.5757) | -202.457 (181.7519) | 273.000 (407.2935) | 1724.197 (901.9847)
  CD206+,Session2,Day3, Pre-fluid sampling,n=2,4,2,4 | -496.500 (422.1427) | -469.550 (397.5609) | -9.500 (504.1671) | 11.054 (268.4708)
  CD209+, Session2,Day1, 40 minutes, n=2,4,2,4 | 15.800 (109.6016) | 4.001 (37.3132) | -9.700 (200.1112) | -16.194 (23.7386)
  CD209+, Session2,Day1,2 hour 40 minutes, n=2,4,2,4 | -78.650 (39.1030) | -9.406 (15.8402) | -2.650 (9.9702) | -10.000 (17.4401)
  CD209+, Session2,Day1,5 hour 40 minutes, n=2,4,2,4 | 17.350 (123.2487) | -17.622 (25.5632) | -44.250 (85.9135) | 10.936 (32.9481)
  CD209+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD209+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | -7.284 (34.7539)
  CD209+,Session2,Day2,Pre-fluid sampling,n=2,4, 2,4 | 36.450 (150.6845) | -3.732 (32.4741) | 174.850 (143.8962) | 71.592 (146.6326)
  CD209+,Session2,Day3, Pre-fluid sampling,n=2,4,2,4 | -30.630 (180.9203) | -7.759 (29.9928) | 5.850 (122.2588) | 23.752 (61.2399)
  CD40, Session2,Day1, 40 minutes, n=2,4,2,4 | -96.5000 (111.01576) | -36.2400 (53.43955) | 340.0000 (53.74012) | -74.1970 (70.63576)
  CD40, Session2,Day1,2 hour 40 minutes, n=2,4,2,4 | -84.0000 (263.04372) | -34.9520 (59.47287) | -97.0000 (43.84062) | -36.8868 (86.92683)
  CD40, Session2,Day1,5 hour 40 minutes, n=2,4,2,4 | -136.5000 (48.79037) | -3.5480 (23.88276) | -62.0000 (117.37973) | -9.8278 (40.48593)
  CD40, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD40, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | 36.2845 (55.24688)
  CD40, Session2,Day2, Pre-fluid sampling,n=2,4, 2,4 | 29.5000 (86.97413) | 76.4310 (173.35366) | 1.0000 (26.87006) | 87.4498 (34.37912)
  CD40, Session2,Day3, Pre-fluid sampling,n=2, 4,2,4 | -184.5000 (20.50610) | -8.5503 (56.03828) | 1.5000 (218.49600) | -33.4253 (54.35736)
  CD80, Session2,Day1, 40 minutes, n=2, 4,2,4 | -56.0000 (15.55635) | 22.5760 (29.07877) | 151.5000 (36.06245) | -10.8950 (7.78157)
  CD80, Session2,Day1,2 hour 40 minutes, n=2,4,2,4 | -48.5000 (85.55992) | -14.4080 (34.73965) | -43.0000 (4.24264) | -11.1910 (6.58469)
  CD80, Session2,Day1,5 hour 40 minutes, n=2, 4,2,4 | -80.5000 (27.57716) | -28.4175 (31.59217) | -112.9000 (97.43931) | -5.9842 (18.30542)
  CD80, Session2,Day1,9 hour 40 minutes, n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD80, Session2,Day1,9 hour 40 minutes, n=0,0,0,4 |  |  |  | 13.1760 (30.88285)
  CD80,Session2,Day2, Pre-fluid sampling,n=2, 4,2,4 | 46.0000 (7.07107) | 33.8863 (44.87592) | 48.0000 (76.36753) | 51.1900 (44.73616)
  CD80,Session2,Day3, Pre-fluid sampling,n=2, 4,2,4 | 45.5000 (78.48885) | 11.4885 (25.25635) | -5.5000 (21.92031) | 29.5018 (31.07571)
  CD83, Session2,Day1, 40 minutes, n=2, 4,2,4 | -360.500 (676.7012) | -509.522 (743.2824) | 341.000 (1500.4806) | 268.284 (705.8063)
  CD83, Session2,Day1,2 hour 40 minutes, n=2, 4,2,4 | 254.500 (866.2058) | -192.732 (586.9635) | -157.500 (96.8736) | 113.359 (989.9087)
  CD83, Session2,Day1,5 hour 40 minutes, n=2, 4,2,4 | -441.500 (844.9926) | 136.272 (346.4007) | 56.500 (610.2332) | -694.319 (570.1803)
  CD83, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD83, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | 450.242 (1654.9166)
  CD83,Session2,Day2, Pre-fluid sampling,n=2, 4,2,4 | -32.000 (394.5656) | 185.975 (797.3145) | -312.000 (417.1930) | -72.629 (223.2647)
  CD83,Session2,Day3, Pre-fluid sampling,n=2, 4,2,4 | -547.000 (687.3078) | -261.969 (458.2399) | -618.500 (1304.6120) | -461.280 (449.4745)
  CD86+, Session2,Day1, 40 minutes, n=2, 4,2,4 | -93.5000 (17.67767) | -51.3590 (54.09737) | -35.0000 (100.40916) | 22.1330 (58.85301)
  CD86+, Session2,Day1,2 hour 40 minutes, n=2, 4,2,4 | 15.5000 (191.62594) | -80.7150 (36.89354) | -62.5000 (40.30509) | 7.4130 (91.99398)
  CD86+, Session2,Day1,5 hour 40 minutes, n=2, 4,2,4 | -130.0000 (65.05382) | -85.0973 (32.66115) | -11.5000 (183.14066) | -77.6915 (70.58944)
  CD86+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD86+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | -58.9008 (99.84882)
  CD86+,Session2,Day2, Pre-fluid sampling,n=2, 4,2,4 | 32.5000 (88.38835) | 43.1203 (47.48816) | 120.5000 (44.54773) | 27.5388 (55.57075)
  CD86+,Session2,Day3, Pre-fluid sampling,n=2, 4,2,4 | -60.5000 (37.47666) | 20.5612 (21.58116) | 35.5000 (153.44217) | -17.0975 (38.55065)
  HLA-DR, Session2,Day1, 40 minutes, n=2, 4,2,4 | -1701.500 (96.8736) | -3036.438 (1102.3399) | -2247.000 (1572.6055) | -1240.116 (874.3051)
  HLA-DR, Session2,Day1,2 hour 40 minutes, n=2,4,2,4 | -706.000 (1269.9638) | -3133.030 (1601.2468) | -1898.000 (733.9768) | -764.884 (1616.7399)
  HLA-DR, Session2,Day1,5 hour 40 minutes, n=2,4,2,4 | -1452.000 (366.2813) | -2242.108 (1155.9978) | -1296.500 (352.8463) | -126.436 (774.0775)
  HLA-DR, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  HLA-DR, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | 798.182 (1011.1423)
  HLA-DR,Session2,Day2, Pre-fluid sampling,n=2,4,2,4 | -171.000 (835.8002) | 924.615 (1288.5384) | 2717.500 (2687.7129) | 904.203 (1067.6177)
  HLA-DR,Session2,Day3, Pre-fluid sampling,n=2,4,2,4 | -957.500 (514.0666) | -978.224 (661.5084) | -3.000 (612.3545) | -549.404 (673.4385)

31. Secondary Outcome: Part 2: Change From Baseline in Cell Activation Markers by Flow Cytometry on Monocytes in Blood
Description: as for outcome 25
Time Frame: Baseline, Session 2: 40 minutes, 2 hour 40 minutes, 5 hour 40 minutes,9hours 40 minutes on Day 1; Pre-fluid sample on Day 2 and Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Part 1: Change From Baseline in Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blood
Description: Blood samples were collected at indicated time-points for the measurement of activation markers by flow cytometry for dendritic cells in blood. Activation markers included CD16, CD163, CD206, CD209, CD40, CD80, CD83, CD86 and HLA-DR. Latest pre-challenge (LPS or GM-CSF) assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Mean fluorescence intensity
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2
Number analyzed (Participants) | 2 | 4 | 2 | 4
Mean fluorescence intensity
  CD16+, Session2,Day1, 40 minutes, n=2, 4, 2,4 | -1492.500 (1341.3816) | -468.314 (270.9419) | -1418.700 (1089.3687) | -215.981 (31.8638)
  CD16+, Session2,Day1, 2 hour 40 minutes, n=2,4,2,4 | -1561.000 (1359.0592) | -579.984 (235.0820) | -1495.500 (1535.1288) | -118.536 (142.1664)
  CD16+, Session2,Day1, 5 hour 40 minutes, n=2,4,2,4 | -1061.000 (823.0723) | -530.365 (208.1743) | -1334.500 (1035.9114) | 171.104 (275.2637)
  CD16+, Session2,Day1,9 hour 40 minutes,n-0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD16+, Session2,Day1,9 hour 40 minutes,n-0,0,0,4 |  |  |  | 265.065 (334.2355)
  CD16+,Session2,Day2, Pre-fluid sampling, n=2,4,2,4 | 135.500 (446.1844) | 300.333 (432.7904) | 309.500 (436.2849) | 168.661 (115.8827)
  CD16+,Session2,Day3, Pre-fluid sampling, n=2,4,2,4 | -564.500 (536.6940) | 1116.482 (840.6096) | 984.000 (130.1076) | 4.757 (149.9929)
  CD163+, Session2,Day1, 40 minutes, n=2,4,2,4 | 41.0000 (65.05382) | -3.8803 (39.59977) | -160.5000 (152.02796) | 58.3640 (66.82273)
  CD163+, Session2,Day1,2 hour 40 minutes, n=2,4,2,4 | -53.5000 (31.81981) | -28.0153 (33.20632) | -187.5500 (156.34131) | 47.3110 (48.31955)
  CD163+, Session2,Day1,5 hour 40 minutes, n=2,4,2,4 | 28.0000 (87.68124) | 13.7295 (38.55623) | -41.5000 (101.11627) | -12.9720 (77.32898)
  CD163+, Session2,Day1, 9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD163+, Session2,Day1, 9 hour 40 minutes,n=0,0,0,4 |  |  |  | -24.0198 (66.75178)
  CD163+,Session2,Day2, Pre-fluid sampling,n=2,4,2,4 | -35.0000 (35.35534) | 68.9850 (76.56191) | 239.0000 (11.31371) | -19.7730 (57.09070)
  CD163+,Session2,Day3, Pre-fluid sampling,n=2,4,2,4 | 38.0000 (50.91169) | 175.6860 (104.35800) | 88.5000 (27.57716) | -10.6642 (38.84898)
  CD206+, Session2,Day1, 40 minutes, n=2,2,2,4: number analyzed (Participants) | 2 | 2 | 2 | 4
  CD206+, Session2,Day1, 40 minutes, n=2,2,2,4 | -75.000 (130.1076) | -140.156 (160.1010) | 241.000 (22.6274) | 552.855 (259.4200)
  CD206+, Session2,Day1,2 hour 40 minutes, n=2,2,2,4: number analyzed (Participants) | 2 | 2 | 2 | 4
  CD206+, Session2,Day1,2 hour 40 minutes, n=2,2,2,4 | 570.500 (164.7559) | -130.065 (141.4567) | 124.000 (229.1026) | 444.094 (454.3525)
  CD206+, Session2,Day1,5 hour 40 minutes, n=2,2,2,4: number analyzed (Participants) | 2 | 2 | 2 | 4
  CD206+, Session2,Day1,5 hour 40 minutes, n=2,2,2,4 | -54.500 (106.7731) | -84.217 (161.6658) | 0.500 (215.6676) | 262.268 (126.1299)
  CD206+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD206+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | 275.423 (163.9991)
  CD206+,Session2,Day2, Pre-fluid sampling,n=2,2,2,4: number analyzed (Participants) | 2 | 2 | 2 | 4
  CD206+,Session2,Day2, Pre-fluid sampling,n=2,2,2,4 | 8.500 (57.2756) | 70.416 (127.1590) | 193.000 (190.9188) | 164.064 (33.1212)
  CD206+,Session2,Day3, Pre-fluid sampling,n=2,2,2,4: number analyzed (Participants) | 2 | 2 | 2 | 4
  CD206+,Session2,Day3, Pre-fluid sampling,n=2,2,2,4 | -87.500 (89.8026) | -7.138 (143.0385) | 120.000 (277.1859) | 106.723 (28.9729)
  CD209+, Session2,Day1, 40 minutes, n=2,4,2,4 | -46.5000 (82.73149) | 18.4320 (55.78181) | -105.6500 (125.08719) | -6.6660 (43.24876)
  CD209+, Session2,Day1,2 hour 40 minutes, n=2,4,2,4 | -42.0000 (16.97056) | -19.1610 (8.85490) | 226.5000 (201.52543) | -19.5825 (32.92128)
  CD209+, Session2,Day1,5 hour 40 minutes, n=2,4,2,4 | -53.5000 (28.99138) | -3.8503 (17.48560) | -42.8500 (1.90919) | -15.8723 (25.15864)
  CD209+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD209+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | -45.1118 (38.63888)
  CD209+,Session2,Day2,Pre-fluid sampling,n=2,4, 2,4 | 6.5000 (53.03301) | -4.8983 (19.52432) | 158.5000 (65.76093) | 46.9815 (100.06420)
  CD209+,Session2,Day3, Pre-fluid sampling,n=2,4,2,4 | -64.5000 (68.58936) | -16.7770 (8.10389) | -9.5000 (58.68986) | -6.7250 (35.83716)
  CD40, Session2,Day1, 40 minutes, n=2,4,2,4 | -77.5000 (105.35891) | 24.1702 (96.21606) | -17.1500 (143.04770) | -37.4720 (29.71510)
  CD40, Session2,Day1,2 hour 40 minutes, n=2,4,2,4 | -248.5000 (194.45436) | -37.2498 (30.55431) | -74.1500 (35.14321) | -11.0400 (65.99710)
  CD40, Session2,Day1,5 hour 40 minutes, n=2,4,2,4 | -191.0000 (22.62742) | -35.5593 (26.02435) | -55.0500 (114.62201) | 78.3045 (54.05275)
  CD40, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD40, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | 102.0438 (67.79389)
  CD40, Session2,Day2, Pre-fluid sampling,n=2,4, 2,4 | -93.0000 (70.71068) | 62.5378 (130.98543) | 135.5000 (51.61880) | 83.1860 (92.90385)
  CD40, Session2,Day3, Pre-fluid sampling,n=2, 4,2,4 | -359.9500 (219.13239) | 108.3750 (91.11295) | 152.5000 (78.48885) | 5.2222 (66.38351)
  CD80, Session2,Day1, 40 minutes, n=2, 4,2,4 | -4.000 (72.1249) | -35.839 (78.4625) | 666.250 (1446.3869) | -11.569 (10.9548)
  CD80, Session2,Day1,2 hour 40 minutes, n=2,4,2,4 | -104.500 (2.1213) | -95.364 (66.7035) | -138.800 (45.5377) | -15.964 (41.2839)
  CD80, Session2,Day1,5 hour 40 minutes, n=2, 4,2,4 | -146.000 (7.0711) | -85.528 (66.3639) | -139.800 (25.7387) | 22.829 (39.2596)
  CD80, Session2,Day1,9 hour 40 minutes, n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD80, Session2,Day1,9 hour 40 minutes, n=0,0,0,4 |  |  |  | 19.214 (43.1702)
  CD80,Session2,Day2, Pre-fluid sampling,n=2, 4,2,4 | 34.000 (31.1127) | 11.103 (88.5547) | 75.000 (26.8701) | 36.587 (15.1919)
  CD80,Session2,Day3, Pre-fluid sampling,n=2, 4,2,4 | -47.500 (2.1213) | 82.987 (84.8958) | 113.500 (16.2635) | 11.929 (20.6629)
  CD83, Session2,Day1, 40 minutes, n=2, 4,2,4 | -225.000 (31.1127) | 0.262 (93.0741) | 647.500 (358.5031) | 8.260 (38.7864)
  CD83, Session2,Day1,2 hour 40 minutes, n=2, 4,2,4 | -26.500 (246.7803) | -56.590 (73.5714) | -17.500 (309.0057) | 4.970 (118.6525)
  CD83, Session2,Day1,5 hour 40 minutes, n=2, 4,2,4 | -127.000 (97.5807) | -54.265 (56.5138) | -40.000 (52.3259) | -11.648 (63.0964)
  CD83, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD83, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | 223.093 (184.1060)
  CD83,Session2,Day2, Pre-fluid sampling,n=2, 4,2,4 | -58.000 (134.3503) | 125.239 (117.8095) | 243.500 (153.4422) | 72.982 (123.0727)
  CD83,Session2,Day3, Pre-fluid sampling,n=2, 4,2,4 | -241.500 (103.9447) | 142.101 (59.5839) | 38.500 (188.7975) | -33.869 (79.7178)
  CD86+, Session2,Day1, 40 minutes, n=2, 4,2,4 | -93.5000 (21.92031) | -101.1600 (78.03703) | 56.0000 (29.69848) | 8.9678 (29.25980)
  CD86+, Session2,Day1,2 hour 40 minutes, n=2, 4,2,4 | 14.0000 (250.31580) | -121.3668 (68.34453) | -144.5000 (28.99138) | 30.0005 (101.61342)
  CD86+, Session2,Day1,5 hour 40 minutes, n=2, 4,2,4 | -54.5000 (40.30509) | -94.3938 (35.37430) | -44.0000 (214.96046) | 106.9465 (53.12949)
  CD86+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  CD86+, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | 118.6338 (49.28502)
  CD86+,Session2,Day2, Pre-fluid sampling,n=2, 4,2,4 | 41.5000 (75.66043) | 126.1853 (105.91022) | 194.5000 (13.43503) | 83.4098 (63.12670)
  CD86+,Session2,Day3, Pre-fluid sampling,n=2, 4,2,4 | -91.0000 (32.52691) | 117.9230 (55.75943) | 82.0000 (94.75231) | 15.2970 (75.45627)
  HLA-DR, Session2,Day1, 40 minutes, n=2, 4,2,4 | 445.50 (434.871) | 896.74 (1309.134) | 41096.00 (47912.141) | -2795.55 (2243.871)
  HLA-DR, Session2,Day1,2 hour 40 minutes, n=2,4,2,4 | -2457.50 (775.696) | -1417.49 (1937.407) | -5430.00 (5929.797) | -1430.37 (2743.193)
  HLA-DR, Session2,Day1,5 hour 40 minutes, n=2,4,2,4 | -320.00 (523.259) | -1744.11 (2077.874) | -1604.00 (3859.389) | -1347.06 (2935.540)
  HLA-DR, Session2,Day1,9 hour 40 minutes,n=0,0,0,4: number analyzed (Participants) | 0 | 0 | 0 | 4
  HLA-DR, Session2,Day1,9 hour 40 minutes,n=0,0,0,4 |  |  |  | -943.38 (4035.982)
  HLA-DR,Session2,Day2, Pre-fluid sampling,n=2,4,2,4 | -1449.00 (1571.191) | 688.02 (1710.854) | -2085.00 (4775.799) | 800.49 (2738.323)
  HLA-DR,Session2,Day3, Pre-fluid sampling,n=2,4,2,4 | -2292.50 (416.486) | -2030.80 (2398.091) | -6379.00 (9237.643) | 113.79 (2769.699)

33. Secondary Outcome: Part 2: Change From Baseline in Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blood
Description: as for outcome 25
Time Frame: as for outcome 5
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Part 1: Change From Baseline in Circulating Leukocyte Numbers in Blood: LPS Arm
Description: Blood samples were collected at indicated time-points for analysis of leukocyte. Latest pre-challenge assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Time Frame: Baseline; Session 2: 40 minutes, 2 hours 40 minutes, 5 hours 40 minutes on Day 1. Pre-fluid sample on Day 2 and Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Cells per milliliter
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg
Number analyzed (Participants) | 2 | 4 | 2
Cells per milliliter
  Session2, Day 1, 40 minutes | -358893.71 (1002862.023) | -1477705.00 (811560.729) | -2065961.83 (1083290.576)
  Session2, Day 1, 2 hours 40 minutes | 3347754.14 (1701524.775) | 2423233.00 (2047535.993) | 5224467.23 (800613.402)
  Session2, Day 1, 5 hours 40 minutes | 2116748.36 (3209541.020) | 4511414.25 (3044446.191) | 3641780.22 (1458532.473)
  Session2, Day 2, Pre-fluid sample | -447452.27 (101410.586) | 881299.75 (1640158.830) | 442226.68 (232936.722)
  Session2, Day 3, Pre-fluid sample | -169328.51 (21593.240) | -93685.25 (1383413.608) | 75348.31 (927892.867)

35. Secondary Outcome: Part 2: Change From Baseline in Circulating Leukocyte Numbers in Blood: LPS Arm
Description: Blood samples were planned to be collected at indicated time-points for the measurement of activation. Latest pre-challenge assessment with a non-missing value, including those from unscheduled visits was considered as Baseline. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Time Frame: Baseline; Session 2: 40 minutes, 2 hours 40 minutes, 5 hours 40 minutes on Day 1. Pre-fluid sample on Day 2 and Day 3
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With LPS
Number analyzed (Participants) | 0

36. Primary Outcome: Part 2: Change From Baseline in White Blood Cell Numbers in Blood: GM-CSF
Description: Blood samples were planned to be collected at indicated time-points for analysis of white blood cells. Baseline value is Session 2 Day 1. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Part 2 of the study was not conducted as agreed criteria for Interim analysis was achieved.
Time Frame: as for outcome 5
Population: Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 2: Participants With GM-CSF
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from the start of study treatment until 69 days in Part 1 of the study.
Description: AEs and SAEs were collected in Part 1 for Safety Population. Data was not collected for Part 2 as participants were not enrolled for Part 2.
Arm/Group | Part 1: LPS 0.5 ng/kg | Part 1: LPS 0.75 ng/kg | Part 1: LPS 1 ng/kg | Part 1: GM-CSF 60 µg/m^2 | Part 2: Participants With LPS | Part 2: Participants With GM-CSF
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/2 | 0/4 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/2 | 0/4 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 2/2 | 3/4 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: LPS 0.5 ng/kg (N=2) | Part 1: LPS 0.75 ng/kg (N=4) | Part 1: LPS 1 ng/kg (N=2) | Part 1: GM-CSF 60 µg/m^2 (N=4) | Part 2: Participants With LPS (N=0) | Part 2: Participants With GM-CSF (N=0)
Chills (General disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT03306589/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT03306589/SAP_001.pdf